CLINICAL TRIAL: NCT02383407
Title: Low Frequency Electrical Stimulation of the Fornix in Intractable Mesial Temporal Lobe Epilepsy (MTLE)
Acronym: MTLE-DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Mohamad Koubeissi, MD, PI, George Washington University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 111239
Record Dates: First submitted 2015-02-19; First posted 2015-03-09 (Estimated); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Mesial Temporal Lobe Epilepsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stimulation group 2 Hz (Experimental): Patient will be randomized to a stimulation group of 2 Hz using Medtronic deep brain stimulation device
  Interventions: Device: Medtronic Deep Brain Stimulation
- Stimulation group 5 Hz (Experimental): Patient will be randomized to a stimulation group of 5 Hz using Medtronic deep brain stimulation device
  Interventions: Device: Medtronic Deep Brain Stimulation

INTERVENTIONS:
Device: Medtronic Deep Brain Stimulation

SUMMARY:
The primary aim of the current proposal is to evaluate safety and tolerability, in terms of neuropsychological effects of low frequency electrical stimulation of the fornix (LFSF) in participants with medically-intractable Mesial Temporal Lobe Epilepsy. Secondary aims include evaluation of psychiatric changes, seizure frequency, and quality of life during LFSF.

DETAILED DESCRIPTION:
Low frequency stimulation is an attractive, uninvestigated method for treatment of intractable epilepsy. Preliminary animal and human data suggest safety and remarkable efficacy of Low frequency stimulation (LFS) in epilepsy. In addition, the duty cycle of LFS is very low, implying less electric current injection, with less charge density on the target tissue and electrodes, and longer battery life. The current project is a classic translational, single-blinded, randomized research project, demonstrating a clear path from the laboratory to bedside. If successful, this new therapy will be of great value to patients with medically and surgically intractable Mesial Temporal Lobe Epilepsy (MTLE).

The study is expected to last approximately 5 years, from enrollment of the first patient to completion of the final subject, taking into consideration attrition and otherwise-eligible subjects who will not elect to participate. Once the study is completed, and enrolled participants have completed all required elements of the protocol, a final report will be submitted to the FDA. Participants may also discontinue their participation in the study, if they wish, at any time.

ELIGIBILITY:
Inclusion Criteria:

* Participants are between the ages of 18 -65 years of age
* Participants must have had a non-invasive video-EEG monitoring revealing seizure semiology and ictal EEG consistent with unilateral or bilateral MTLE
* Participants must have tried and failed two trials of antiepileptic drugs (AEDs)
* Participants may have lesional or non lesional hippocampi, as evidenced by brain MRI acquired within the previous two years
* Participants are prescribed and taking 1-4 AEDs at the time of study entry
* Study participants will have intractable (MTLE) with a seizure frequency of at least 1/month averaged over the preceding 6 months prior to enrollment, including maximum seizure-freedom periods of no more than 60 days.
* Participants must have a platelet count greater than 125,000 per cubic millimeter and prothrombin time (PT) and activated partial thromboplastin time (aPTT) within normal limits at the visit prior to surgery

Exclusion Criteria:

* Progressive neurological or medical diseases, such as brain tumors or neurodegenerative disease or cancer
* Non-compliance with antiepileptic medications as demonstrated by the medical record
* Any conditions interfering with electrode implantation
* Any non-epileptic seizures
* Inability or unwillingness to complete neuropsychological tests or complete seizure diaries
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Pregnant, or planning to become pregnant*
* Participation in another research trial where the participant was treated with another investigational drug or device within 30 days prior to enrollment of study
* Intelligence Quotient showing a general ability Quotient of less than 70. The score excludes the contribution of working memory and processing speed (which are areas of cognitive functioning that are vulnerable to numerous influences including seizures and fatigue and effects of AEDs)
* Inability or unwillingness of individual to give written informed consent
* Participants who have changes to their antiepileptic medications during the baseline phase (as they will need to repeat the baseline phase)
* Subjects with history of status epilepticus within the preceding year
* History of psychiatric illness necessitating hospitalizations
* Subjects who have any of the following implanted devices: aneurysm clips, cardiac pacemaker or defibrillator, cochlear implant, spinal cord, DBS, or vagal nerve stimulator
* Co-morbid conditions that would interfere with study stimulation activities or response to treatment, which may include:

  * Neoplasm with life expectancy < 5 years
  * Severe chronic pulmonary disease
  * Local, systemic acute or chronic infectious illness
  * Life threatening cardiac arrhythmias
  * Severe collagen vascular disorder
  * Kidney failure or other major organ system failures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-12; Primary Completion 2018-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GW Medical Faculty Associates, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Koubeissi MZ, Joshi S, Eid A, Emami M, Jaafar N, Syed T, Foreman PJ, Sheth A, Amdur R, Bou Nasif M, Puente AN, Aly R, Chen H, Becker A, Gholipour T, Makke Y, Elmashad A, Gagnon L, Durand DM, Gaillard WD, Shields DC. Low-frequency stimulation of a fiber tract in bilateral temporal lobe epilepsy. Epilepsy Behav. 2022 May;130:108667. doi: 10.1016/j.yebeh.2022.108667. Epub 2022 Mar 26. PMID 35344808
- See also: PubMed — https://pubmed.ncbi.nlm.nih.gov/35344808/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Once screened and enrolled, all subjects underwent implantation of SEEG electrodes in both hippocampi orthogonally through the lateral temporal neocortex. 2 patients were excluded as one opted for temporal lobectomy, and the other for multiple hippocampal transections. The implanted subjects did not receive stimulation for 1-month postoperatively then were randomized to either 2-Hz or 5-Hz.
Groups:
- Stimulation Group 2 Hz: Patient will be randomized to a stimulation group of 2 Hz using Medtronic deep brain stimulation device
  Medtronic Deep Brain Stimulation
- Stimulation Group 5 Hz: Patient will be randomized to a stimulation group of 5 Hz using Medtronic deep brain stimulation device
  Medtronic Deep Brain Stimulation
Period: Overall Study
Arm/Group | Stimulation Group 2 Hz | Stimulation Group 5 Hz
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2 Hz: Patient will be randomized to a stimulation group of 2 Hz using Medtronic deep brain stimulation device
- 5 Hz: Patient will be randomized to a stimulation group of 5 Hz using Medtronic deep brain stimulation device
- Total: Total of all reporting groups
Arm/Group | 2 Hz | 5 Hz | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 36 [36 to 36] | 46 [46 to 46] | 42.7 [36 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Bilateral temporal lobe epilepsy [Count of Participants; unit: Participants] | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Low Frequency Stimulation of the Fornix With Regards to Memory Function
Description: The primary outcome is safety and tolerability of LFSF in participants with intractable MTLE with regards to memory function. The number of participants listed are those who had a significant changes in RAVLT score.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 2 Hz | 5 Hz
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

2. Secondary Outcome: Psychiatric Health (Effects of LFS on Psychiatric Symptoms Using Standardized Measures That Are Known to be Sensitive to Changes to Surgical Treatment of TLE)
Description: Since LFSF is expected to activate limbic structures, we will assess the effects of LFS on psychiatric symptoms using standardized measures that are known to be sensitive to changes to surgical treatment of TLE. The number of participation listed are those who had a significant change in anxiety, depression, or suicidality based on a qualitative overview of the psychiatric assessments performed preoperatively and postoperatively.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 2 Hz | 5 Hz
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

3. Secondary Outcome: To Assess if Electrode Implantation in the Fornix is Feasible as is Done in Patients With Parkinson's Disease.
Description: The DBS leads are routinely implanted for patients with Parkinson's disease. Thus, we planned to implant Model 3389 DBS leads using the same technique of stereotactic implantation. A secondary aim of this trial is to standardize the implantation, the evoked potential and electric current determination procedures in preparation for a large-scale phase III trial. The number of participants with the outcome measure are those in whom bilateral hippocampal CCEPs were consistently present.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 2 Hz | 5 Hz
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

4. Secondary Outcome: Effect on Seizure Frequency
Description: Seizure reduction: Subjects underwent implantation of pulse generators and long-term low-frequency stimulation with mean monthly seizures during blinded phase
Time Frame: 1 year
Population: arms were combined for safety reasons.
Measure: Mean (Standard Deviation); unit: Seizure per week
Groups:
- Stimulation on: Both arms analyzed with the DBS stimulation on (frequency of 5 Hz)
- Stimulation Off: Both arms analyzed with the DBS stimulation off (frequency of 5 Hz)
Arm/Group | Stimulation on | Stimulation Off
Number analyzed (Participants) | 3 | 3
Seizure per week | 0.96 (1.23) | 3.14 (2.67)

5. Secondary Outcome: Effect on Seizure Frequency
Description: as for outcome 4
Time Frame: 1 year
Population: arms were combined for safety reasons.
Measure: Mean (Standard Deviation); unit: Seizure per week
Groups:
- Stimulation on: Both arms analyzed with the DBS stimulation on (frequency of 2 Hz)
- Stimulation Off: Both arms analyzed with the DBS stimulation off (frequency of 2 Hz)
Arm/Group | Stimulation on | Stimulation Off
Number analyzed (Participants) | 3 | 3
Seizure per week | 0.96 (1.23) | 3.14 (2.67)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded at each follow up visit, after implantation of the divide, follow-up was every 2 months for 12 months, then less regularly during the post blinding period for 12 months. Participants also reached out directly to the team between follow ups if they were to have any adverse events.
Description: Adverse events were recorded at each follow up visit as detailed above.
Arm/Group | 2 Hz | 5 Hz
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 Hz (N=1) | 5 Hz (N=2)
Intraparenchymal hemorrhage (Nervous system disorders) | 0 | 1 (1) — ICU admission for sudden onset of aphasia due to intraparenchymal hemorrhage in the left temporal lobe. Patient discharged with anomia and verbal memory deficits, gradually improved. The DSMB deemed the hemorrhage unrelated to the DBS implantation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT02383407/Prot_SAP_000.pdf
  • Informed Consent Form (2015-12-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT02383407/ICF_001.pdf